CLINICAL TRIAL: NCT01943825
Title: Exploration of Immunologic Mechanisms of Immune Interference and/or Cross-Neutralizing Immunity Following Various Administration Schedules With CYD Tetravalent Dengue Vaccine
Brief Title: Immunologic Mechanisms of Immune Interference and/or Cross-Neutralizing Immunity After CYD Tetravalent Dengue Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD56; U1111-1143-8391 (Other: WHO)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue; Dengue fever; CYD dengue vaccine; IXIARO JE vaccine; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CYD Dengue Vaccine: Group 1 (Experimental): Participants received 3 doses of CYD dengue vaccine, one each at 0, 2 and 6 months, respectively.
  Interventions: Biological: CYD Dengue Vaccine
- CYD Dengue Vaccine: Group 2 (Experimental): Participants received 3 doses of CYD dengue vaccine, one each at 0, 6 and 12 months, respectively.
  Interventions: Biological: CYD Dengue Vaccine
- CYD Dengue and JE Vaccine: Group 3 (Experimental): Participants received 3 doses of CYD dengue vaccine, one each at 0, 2 and 6 months, and 2 doses of JE (IXIARO) vaccine at 0 and 1 months, respectively.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Japanese Encephalitis Vaccine
- CYD Dengue and JE Vaccine: Group 4 (Experimental): Participants received 2 doses of JE (IXIARO) vaccine at 0 and 1 months; and 3 doses of CYD dengue vaccine at 7, 9 and 13 months, respectively.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Japanese Encephalitis Vaccine

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous
  Arms: CYD Dengue Vaccine: Group 1; CYD Dengue and JE Vaccine: Group 3; CYD Dengue and JE Vaccine: Group 4
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous
  Arms: CYD Dengue Vaccine: Group 2
Biological: Japanese Encephalitis Vaccine — 0.5 mL, Intramuscular
  Other Names: IXIARO Japanese Encephalitis Vaccine
  Arms: CYD Dengue and JE Vaccine: Group 3
Biological: Japanese Encephalitis Vaccine — 0.5 mL, Intramuscular
  Other Names: IXIARO Japanese Encephalitis Vaccine
  Arms: CYD Dengue and JE Vaccine: Group 4

SUMMARY:
The aim of the study was to evaluate a compressed dosing schedule and the immunologic effects of co-administration of a CYD dengue vaccine with a licensed flavivirus (FV) with Japanese encephalitis (JE) vaccine.

Primary Objectives:

* To describe and compare the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after each CYD dengue vaccine dose.
* To describe the persistence of the humoral immune response to each of the 4 parental dengue virus serotypes 6 after CYD dengue vaccine Dose 3, irrespective of whether or not JE vaccine had been previously administered.

Secondary Objectives:

* To describe the safety profile after each injection of CYD dengue vaccine.
* To describe the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after each CYD dengue vaccine dose when administered with or after JE virus vaccine in Groups 3 and 4.
* To describe the persistence of the humoral immune response to each of the 4 parental dengue virus serotypes at 6 months post-dose 3 in all four groups and at 12 months post-dose 3 in Groups 1 and 3 with the compressed schedule.
* To determine the level of viremia on Day (D)0, D3, D5, D7 and D14 following each CYD vaccine dose administered in Groups 1-4.
* To describe the JE humoral immune response at baseline and 28 days after each injection of CYD dengue vaccine in Groups 3 and 4.

DETAILED DESCRIPTION:
Study participants were randomly assigned to one of the four groups to receive assigned study vaccine and were evaluated for neutralizing antibody titers; markers of cell-mediated immunity.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to (>=)18 to less than or equal to (<=) 45 years on the day of inclusion.
* Informed consent form had been signed and dated.
* Able to attend all scheduled visits and complied with all trial procedures.
* Participant was in good health, based on medical history and physical examination.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (were considered of non-childbearing potential, a female had to be post- menopausal for at least 1 year, surgically sterile, or used an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
* Participation in the 4 weeks preceding the first trial vaccination, or planned participation during the present trial period, in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt or planned receipt of any vaccine, outside the study protocol in the 4 weeks preceded or followed trial vaccinations. (If influenza activity warranted vaccination of healthy young adults, influenza vaccination was encouraged and did not lead to study exclusion).
* Any history of FV vaccination, or planned FV vaccination during the trial period.
* Previous residence (greater than [>]12 months) in, or travel in the last 30 days to dengue endemic regions.
* Receipt of immune globulins, blood or blood-derived products in the 3 months prior to first vaccination or planned use during the study period.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceded 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components (including protamine sulfate), or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances, including dry natural latex.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Excessive alcohol consumption or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Identified as an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employee or the Investigator.
* Temporary Exclusion Criteria: Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [>= 100.4 degree fahrenheit]). A prospective participant was not included in the study until the condition had resolved or the febrile event had subsided. If the delay for the febrile illness exceeded the window between screening and vaccination, or if deemed necessary by the Investigator, a prospective participant might be re-screened once the fever had resolved.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were involved in the study from 05 November 2013 to 25 November 2015 in the United States.
Pre-assignment Details: A total of 90 participants were enrolled and randomized in the study.
Groups:
- CYD Dengue and Japanese Encephalitis (JE) Vaccine : Group 3: Participants received 3 doses of CYD dengue vaccine, one each at 0, 2 and 6 months, and 2 doses of JE (IXIARO) vaccine at 0 and 1 months, respectively.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Japanese Encephalitis (JE) Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Started | 25 | 15 | 25 | 25
Completed | 15 | 11 | 10 | 14
Not Completed | 10 | 4 | 15 | 11
Not completed — Lost to Follow-up | 9 | 3 | 12 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 2
Not completed — Other than specified above | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set which included all participants who received at least one dose of CYD dengue vaccine or JE vaccine.
Groups:
- CYD Dengue and JE Vaccine : Group 3: Participants received 3 doses of CYD dengue vaccine, one each at 0, 2 and 6 months, and 2 doses of JE (IXIARO) vaccine at 0 and 1 months, respectively.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4 | Total
Number analyzed (Participants) | 25 | 15 | 25 | 25 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (6.7) | 26.8 (5.6) | 28.5 (6.5) | 30.4 (6.2) | 29.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 7 | 12 | 37
  Male | 13 | 9 | 18 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: Geometric Means Titers (GMTs) of Antibodies Against Each Dengue Virus Serotype Strains
Description: GMTs of antibodies against each dengue virus serotype (parental strains 1, 2, 3 and 4) were measured by plaque reduction neutralization test (PRNT). The lower limit of quantitation (LLOQ) of the assay was a titer of 10 (1/dilution).
Time Frame: Pre-injection 1, 2 and 3; 28 days post-injection 1, 2 and 3; and 6 months post-injection 3
Population: Analysis was performed on full analysis set which included participants who received at least one injection of CYD dengue vaccine or JE vaccine and had at least one blood sample drawn and valid post-injection serology result. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 15 | 25 | 25
titers (1/dilution)
  Serotype 1: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 1: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as less than (<) LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 1: 28 days Post-injection 1 | 6.1 [4.8 to 7.8] | 5.5 [4.5 to 6.8] | 6.8 [4.7 to 10.0] | 7.4 [5.3 to 10.2]
  Serotype 1: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 1: Pre-injection 2 | 6.5 [4.7 to 8.9] | 5.4 [4.6 to 6.4] | 6.7 [4.3 to 10.6] | 7.2 [5.0 to 10.2]
  Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 1: 28 days Post-injection 2 | 8.5 [5.5 to 13.1] | 6.2 [4.5 to 8.4] | 10.8 [5.4 to 21.8] | 10.8 [6.6 to 17.7]
  Serotype 1: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 1: Pre-injection 3 | 7.1 [4.7 to 10.8] | 6.3 [4.4 to 9.0] | 8.3 [4.6 to 15.1] | 6.5 [4.7 to 9.1]
  Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 1: 28 days Post-injection 3 | 9.1 [5.5 to 15.0] | 9.9 [6.0 to 16.6] | 12.0 [5.4 to 26.7] | 12.9 [7.6 to 21.9]
  Serotype 1: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 1: 6 months Post-injection 3 | 5.8 [4.7 to 7.3] | 6.6 [4.3 to 9.9] | 8.6 [3.5 to 21.1] | 7.3 [5.0 to 10.9]
  Serotype 2: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 2: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 2: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 2: 28 days Post-injection 1 | 9.2 [5.3 to 16.1] | 7.4 [4.1 to 13.1] | 8.8 [5.0 to 15.6] | 35.5 [21.2 to 59.5]
  Serotype 2: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 2: Pre-injection 2 | 12.1 [5.3 to 27.4] | 9.6 [5.8 to 15.9] | 8.8 [4.8 to 16.1] | 44.5 [23.1 to 85.7]
  Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 2: 28 days Post-injection 2 | 19.0 [8.8 to 41.1] | 10.7 [5.7 to 19.9] | 17.3 [7.6 to 39.7] | 61.5 [30.4 to 124.6]
  Serotype 2: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 2: Pre-injection 3 | 13.3 [6.7 to 26.4] | 9.8 [5.1 to 18.8] | 12.2 [6.7 to 22.2] | 37.4 [16.1 to 87.1]
  Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 2: 28 days Post-injection 3 | 32.5 [14.3 to 73.9] | 25.5 [13.0 to 50.0] | 19.3 [9.8 to 37.9] | 48.2 [22.4 to 103.5]
  Serotype 2: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 2: 6 months Post-injection 3 | 13.9 [6.7 to 29.0] | 7.9 [4.4 to 14.3] | 10.9 [4.6 to 26.0] | 21.0 [9.2 to 48.2]
  Serotype 3: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 3: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | 5.2 [4.8 to 5.6] | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 3: 28 days Post-injection 1 | 22.1 [12.1 to 40.5] | 24.9 [8.5 to 72.9] | 19.7 [8.8 to 44.1] | 49.3 [24.9 to 97.5]
  Serotype 3: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 3: Pre-injection 2 | 24.5 [10.7 to 56.4] | 15.4 [7.5 to 31.6] | 23.8 [10.8 to 52.4] | 49.0 [22.9 to 104.8]
  Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 3: 28 days Post-injection 2 | 31.0 [15.0 to 63.7] | 40.8 [14.7 to 113.3] | 28.5 [12.4 to 65.4] | 68.8 [36.9 to 128.3]
  Serotype 3: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 3: Pre-injection 3 | 22.9 [12.1 to 43.2] | 31.7 [13.9 to 72.0] | 20.5 [9.5 to 44.1] | 35.6 [17.8 to 71.6]
  Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 3: 28 days Post-injection 3 | 45.5 [24.4 to 84.8] | 79.9 [44.1 to 144.6] | 32.2 [12.9 to 80.7] | 61.8 [39.3 to 97.1]
  Serotype 3: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 3: 6 months Post-injection 3 | 19.3 [10.2 to 36.6] | 33.9 [13.9 to 82.5] | 19.3 [7.5 to 49.5] | 24.8 [12.6 to 48.7]
  Serotype 4: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 4: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 4: 28 days Post-injection 1 | 425.8 [172.1 to 1053.4] | 669.7 [188.3 to 2381.8] | 177.6 [62.1 to 508.1] | 325.4 [147.8 to 716.3]
  Serotype 4: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 4: Pre-injection 2 | 296.2 [151.9 to 577.6] | 100.3 [51.7 to 194.6] | 89.9 [24.8 to 326.2] | 300.9 [144.4 to 627.0]
  Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 4: 28 days Post-injection 2 | 166.6 [90.2 to 307.7] | 147.1 [91.8 to 235.7] | 68.0 [23.4 to 197.1] | 211.3 [103.3 to 432.2]
  Serotype 4: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 4: Pre-injection 3 | 108.9 [63.5 to 186.6] | 89.8 [49.2 to 163.9] | 47.7 [18.4 to 123.9] | 139.5 [65.8 to 295.4]
  Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 4: 28 days Post-injection 3 | 120.4 [67.2 to 215.7] | 124.5 [78.2 to 198.1] | 55.4 [22.5 to 136.8] | 152.5 [75.3 to 308.6]
  Serotype 4: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 4: 6 months Post-injection 3 | 105.3 [52.5 to 211.1] | 106.7 [71.7 to 158.8] | 43.8 [13.3 to 144.3] | 92.6 [56.7 to 151.1]

2. Primary Outcome: Number of Participants With Antibody Titers Greater Than or Equal to (>=)10 (1/Dilution) Against Each Dengue Virus Serotype Strains
Description: Antibody titers against each dengue virus serotype (parental strains 1, 2, 3 and 4) were measured by PRNT.
Time Frame: Pre-injection 1, 2 and 3; 28 days post-injection 1, 2 and 3; and 6 months post-injection 3
Population: Analysis was performed on full analysis set. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Groups:
- CYD Dengue and JE Vaccine : Group 3: Participants received 3 doses of CYD dengue vaccine, one each at 0, 2 and 6 months, and 2 doses of JE (IXIARO) vaccines at 0 and 1 months, respectively.
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 15 | 25 | 25
Participants
  Serotype 1: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 1: Pre-injection 1 | 0 | 0 | 0 | 0
  Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 1: 28 days Post-injection 1 | 3 | 1 | 3 | 6
  Serotype 1: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 1: Pre-injection 2 | 3 | 1 | 2 | 4
  Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 1: 28 days Post-injection 2 | 6 | 2 | 5 | 8
  Serotype 1: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 1: Pre-injection 3 | 3 | 2 | 3 | 3
  Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 1: 28 days Post-injection 3 | 5 | 6 | 5 | 9
  Serotype 1: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 1: 6 months Post-injection 3 | 2 | 2 | 2 | 4
  Serotype 2: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 2: Pre-injection 1 | 0 | 0 | 0 | 0
  Serotype 2: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 2: 28 days Post-injection 1 | 5 | 2 | 4 | 16
  Serotype 2: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 2: Pre-injection 2 | 5 | 7 | 4 | 15
  Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 2: 28 days Post-injection 2 | 9 | 5 | 7 | 16
  Serotype 2: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 2: Pre-injection 3 | 8 | 4 | 7 | 13
  Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 2: 28 days Post-injection 3 | 12 | 9 | 9 | 15
  Serotype 2: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 2: 6 months Post-injection 3 | 7 | 3 | 4 | 9
  Serotype 3: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 3: Pre-injection 1 | 0 | 0 | 1 | 0
  Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 3: 28 days Post-injection 1 | 15 | 7 | 10 | 16
  Serotype 3: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 3: Pre-injection 2 | 11 | 7 | 10 | 14
  Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 3: 28 days Post-injection 2 | 12 | 9 | 10 | 16
  Serotype 3: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 3: Pre-injection 3 | 12 | 10 | 9 | 12
  Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 3: 28 days Post-injection 3 | 14 | 12 | 9 | 16
  Serotype 3: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 3: 6 months Post-injection 3 | 10 | 9 | 6 | 10
  Serotype 4: Pre-injection 1: number analyzed (Participants) | 25 | 15 | 25 | 19
  Serotype 4: Pre-injection 1 | 0 | 0 | 0 | 0
  Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 24 | 14 | 19 | 19
  Serotype 4: 28 days Post-injection 1 | 21 | 13 | 16 | 18
  Serotype 4: Pre-injection 2: number analyzed (Participants) | 22 | 14 | 17 | 18
  Serotype 4: Pre-injection 2 | 21 | 13 | 11 | 18
  Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 18 | 13 | 15 | 18
  Serotype 4: 28 days Post-injection 2 | 17 | 13 | 11 | 18
  Serotype 4: Pre-injection 3: number analyzed (Participants) | 18 | 12 | 15 | 16
  Serotype 4: Pre-injection 3 | 17 | 12 | 11 | 16
  Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 17 | 12 | 14 | 16
  Serotype 4: 28 days Post-injection 3 | 16 | 12 | 11 | 16
  Serotype 4: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 4: 6 months Post-injection 3 | 15 | 11 | 7 | 14

3. Secondary Outcome: Geometric Means Titers of Antibodies Against Each Dengue Virus Serotype Strains in Participants Who Received Japanese Encephalitis Vaccine - Groups 3 and 4
Description: GMTs of antibodies against each dengue virus serotype (parental strains 1, 2, 3 and 4) were measured by PRNT. The LLOQ of the assay was a titer of 10 (1/dilution).
Time Frame: Pre-injection 1, 2 and 3, and 28 days post-injection 1, 2 and 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 25
titers (1/dilution)
  Serotype 1: Pre-injection 1: number analyzed (Participants) | 25 | 19
  Serotype 1: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 19 | 19
  Serotype 1: 28 days Post-injection 1 | 6.8 [4.7 to 10.0] | 7.4 [5.3 to 10.2]
  Serotype 1: Pre-injection 2: number analyzed (Participants) | 17 | 18
  Serotype 1: Pre-injection 2 | 6.7 [4.3 to 10.6] | 7.2 [5.0 to 10.2]
  Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 15 | 18
  Serotype 1: 28 days Post-injection 2 | 10.8 [5.4 to 21.8] | 10.8 [6.6 to 17.7]
  Serotype 1: Pre-injection 3: number analyzed (Participants) | 15 | 16
  Serotype 1: Pre-injection 3 | 8.3 [4.6 to 15.1] | 6.5 [4.7 to 9.1]
  Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 14 | 16
  Serotype 1: 28 days Post-injection 3 | 12.0 [5.4 to 26.7] | 12.9 [7.6 to 21.9]
  Serotype 2: Pre-injection 1: number analyzed (Participants) | 25 | 19
  Serotype 2: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 2: 28 days Post-injection 1: number analyzed (Participants) | 19 | 19
  Serotype 2: 28 days Post-injection 1 | 8.8 [5.0 to 15.6] | 35.5 [21.2 to 59.5]
  Serotype 2: Pre-injection 2: number analyzed (Participants) | 17 | 18
  Serotype 2: Pre-injection 2 | 8.8 [4.8 to 16.1] | 44.5 [23.1 to 85.7]
  Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 15 | 18
  Serotype 2: 28 days Post-injection 2 | 17.3 [7.6 to 39.7] | 61.5 [30.4 to 124.6]
  Serotype 2: Pre-injection 3: number analyzed (Participants) | 15 | 16
  Serotype 2: Pre-injection 3 | 12.2 [6.7 to 22.2] | 37.4 [16.1 to 87.1]
  Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 14 | 16
  Serotype 2: 28 days Post-injection 3 | 19.3 [9.8 to 37.9] | 48.2 [22.4 to 103.5]
  Serotype 3: Pre-injection 1: number analyzed (Participants) | 25 | 19
  Serotype 3: Pre-injection 1 | 5.2 [4.8 to 5.6] | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 19 | 19
  Serotype 3: 28 days Post-injection 1 | 19.7 [8.8 to 44.1] | 49.3 [24.9 to 97.5]
  Serotype 3: Pre-injection 2: number analyzed (Participants) | 17 | 18
  Serotype 3: Pre-injection 2 | 23.8 [10.8 to 52.4] | 49.0 [22.9 to 104.8]
  Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 15 | 18
  Serotype 3: 28 days Post-injection 2 | 28.5 [12.4 to 65.4] | 68.8 [36.9 to 128.3]
  Serotype 3: Pre-injection 3: number analyzed (Participants) | 15 | 16
  Serotype 3: Pre-injection 3 | 20.5 [9.5 to 44.1] | 35.6 [17.8 to 71.6]
  Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 14 | 16
  Serotype 3: 28 days Post-injection 3 | 32.2 [12.9 to 80.7] | 61.8 [39.3 to 97.1]
  Serotype 4: Pre-injection 1: number analyzed (Participants) | 25 | 19
  Serotype 4: Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | NA [NA to NA] — Participants had a titer reported as < LLOQ.
  Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 19 | 19
  Serotype 4: 28 days Post-injection 1 | 177.6 [62.1 to 508.1] | 325.4 [147.8 to 716.3]
  Serotype 4: Pre-injection 2: number analyzed (Participants) | 17 | 18
  Serotype 4: Pre-injection 2 | 89.9 [24.8 to 326.2] | 300.9 [144.4 to 627.0]
  Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 15 | 18
  Serotype 4: 28 days Post-injection 2 | 68.0 [23.4 to 197.1] | 211.3 [103.3 to 432.2]
  Serotype 4: Pre-injection 3: number analyzed (Participants) | 15 | 16
  Serotype 4: Pre-injection 3 | 47.7 [18.4 to 123.9] | 139.5 [65.8 to 295.4]
  Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 14 | 16
  Serotype 4: 28 days Post-injection 3 | 55.4 [22.5 to 136.8] | 152.5 [75.3 to 308.6]

4. Secondary Outcome: Geometric Means Titers of Antibodies Against Each Dengue Virus Serotype Strains
Description: GMTs of antibodies against each dengue virus serotype (parental strains 1, 2, 3 and 4) were measured by PRNT.
Time Frame: 6 months and 12 months post-injection 3
Population: Analysis was performed on full analysis set. Here, 'Number analyzed' = participants with available data for each specified category. Data was not planned to be collected and analyzed for Groups 2 and 4 for 12 months post-injection 3 time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 15 | 25 | 25
titers (1/dilution)
  Serotype 1: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 1: 6 months Post-injection 3 | 5.8 [4.7 to 7.3] | 6.6 [4.3 to 9.9] | 8.6 [3.5 to 12.1] | 7.3 [5.0 to 10.9]
  Serotype 2: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 2: 6 months Post-injection 3 | 13.9 [6.7 to 29.0] | 7.9 [4.4 to 14.3] | 10.9 [4.6 to 26.0] | 21.0 [9.2 to 48.2]
  Serotype 3: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 3: 6 months Post-injection 3 | 19.3 [10.2 to 36.6] | 33.9 [13.9 to 82.5] | 19.3 [7.5 to 49.5] | 24.8 [12.6 to 48.7]
  Serotype 4: 6 months Post-injection 3: number analyzed (Participants) | 17 | 11 | 10 | 14
  Serotype 4: 6 months Post-injection 3 | 105.3 [52.5 to 211.1] | 106.7 [71.7 to 158.8] | 43.8 [13.3 to 144.3] | 92.6 [56.7 to 151.1]
  Serotype 1: 12 months Post-injection 3: number analyzed (Participants) | 15 | 0 | 10 | 0
  Serotype 1: 12 months Post-injection 3 | 5.3 [4.7 to 6.0] |  | 7.8 [4.2 to 14.5] |
  Serotype 2: 12 months Post-injection 3: number analyzed (Participants) | 15 | 0 | 10 | 0
  Serotype 2: 12 months Post-injection 3 | 11.5 [5.2 to 25.5] |  | 7.6 [3.7 to 15.6] |
  Serotype 3: 12 months Post-injection 3: number analyzed (Participants) | 15 | 0 | 10 | 0
  Serotype 3: 12 months Post-injection 3 | 18.3 [9.5 to 35.2] |  | 16.2 [5.8 to 45.0] |
  Serotype 4: 12 months Post-injection 3: number analyzed (Participants) | 15 | 0 | 10 | 0
  Serotype 4: 12 months Post-injection 3 | 144.8 [68.8 to 304.8] |  | 23.9 [8.1 to 70.8] |

5. Secondary Outcome: Number of Participants With Detectable Non Serotype-Specific Vaccine Viremia
Description: Viremia was determined by reverse transcriptase (RT) polymerase chain reaction (PCR) using primer/probes specific to a non serotype-specific part of the dengue vaccine.
Time Frame: 3, 5, 7 and 14 days post-injection 1, 2 and 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 15 | 25 | 25
Participants
  3 days Post-Injection 1: number analyzed (Participants) | 24 | 15 | 22 | 19
  3 days Post-Injection 1 | 0 | 0 | 0 | 1
  5 days Post-Injection 1: number analyzed (Participants) | 24 | 15 | 21 | 19
  5 days Post-Injection 1 | 7 | 5 | 1 | 3
  7 days Post-Injection 1: number analyzed (Participants) | 24 | 15 | 20 | 19
  7 days Post-Injection 1 | 16 | 9 | 8 | 9
  14 days Post-Injection 1: number analyzed (Participants) | 23 | 15 | 18 | 19
  14 days Post-Injection 1 | 12 | 4 | 3 | 6
  3 days Post-Injection 2: number analyzed (Participants) | 22 | 14 | 16 | 17
  3 days Post-Injection 2 | 0 | 0 | 0 | 1
  5 days Post-Injection 2: number analyzed (Participants) | 21 | 14 | 17 | 18
  5 days Post-Injection 2 | 0 | 0 | 0 | 0
  7 days Post-Injection 2: number analyzed (Participants) | 20 | 13 | 17 | 18
  7 days Post-Injection 2 | 0 | 0 | 0 | 0
  14 days Post-Injection 2: number analyzed (Participants) | 19 | 14 | 16 | 18
  14 days Post-Injection 2 | 1 | 1 | 0 | 0
  3 days Post-Injection 3: number analyzed (Participants) | 18 | 11 | 15 | 15
  3 days Post-Injection 3 | 0 | 0 | 0 | 0
  5 days Post-Injection 3: number analyzed (Participants) | 17 | 12 | 15 | 16
  5 days Post-Injection 3 | 0 | 0 | 0 | 0
  7 days Post-Injection 3: number analyzed (Participants) | 18 | 12 | 14 | 16
  7 days Post-Injection 3 | 1 | 0 | 0 | 0
  14 days Post-Injection 3: number analyzed (Participants) | 18 | 12 | 14 | 16
  14 days Post-Injection 3 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Detectable Serotype-Specific Vaccine Viremia
Description: Viremia was determined by RT PCR using primer/probes specific to each dengue vaccine serotypes.
Time Frame: 3, 5, 7 and 14 days post-injection 1; 3 and 14 days post-injection 2 and 7 days post-injection 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 15 | 25 | 25
Participants
  Serotype 1: 3 days Post-Injection 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 1: 3 days Post-Injection 1 |  |  |  | 0
  Serotype 1: 5 days Post-Injection 1: number analyzed (Participants) | 7 | 5 | 1 | 3
  Serotype 1: 5 days Post-Injection 1 | 0 | 0 | 0 | 0
  Serotype 1: 7 days Post-Injection 1: number analyzed (Participants) | 16 | 9 | 8 | 9
  Serotype 1: 7 days Post-Injection 1 | 0 | 1 | 0 | 0
  Serotype 1: 14 days Post-Injection 1: number analyzed (Participants) | 12 | 4 | 3 | 6
  Serotype 1: 14 days Post-Injection 1 | 0 | 0 | 0 | 0
  Serotype 1: 3 days Post-Injection 2: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 1: 3 days Post-Injection 2 |  |  |  | 0
  Serotype 1: 14 days Post-Injection 2: number analyzed (Participants) | 1 | 1 | 0 | 0
  Serotype 1: 14 days Post-Injection 2 | 0 | 0 |  |
  Serotype 1: 7 days Post-Injection 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Serotype 1: 7 days Post-Injection 3 | 0 |  |  |
  Serotype 2: 3 days Post-Injection 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 2: 3 days Post-Injection 1 |  |  |  | 0
  Serotype 2: 5 days Post-Injection 1: number analyzed (Participants) | 7 | 5 | 1 | 3
  Serotype 2: 5 days Post-Injection 1 | 2 | 0 | 0 | 0
  Serotype 2: 7 days Post-Injection 1: number analyzed (Participants) | 16 | 9 | 8 | 9
  Serotype 2: 7 days Post-Injection 1 | 2 | 1 | 1 | 0
  Serotype 2: 14 days Post-Injection 1: number analyzed (Participants) | 12 | 4 | 3 | 6
  Serotype 2: 14 days Post-Injection 1 | 1 | 0 | 0 | 0
  Serotype 2: 3 days Post-Injection 2: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 2: 3 days Post-Injection 2 |  |  |  | 0
  Serotype 2: 14 days Post-Injection 2: number analyzed (Participants) | 1 | 1 | 0 | 0
  Serotype 2: 14 days Post-Injection 2 | 0 | 0 |  |
  Serotype 2: 7 days Post-Injection 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Serotype 2: 7 days Post-Injection 3 | 0 |  |  |
  Serotype 3: 3 days Post-Injection 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 3: 3 days Post-Injection 1 |  |  |  | 0
  Serotype 3: 5 days Post-Injection 1: number analyzed (Participants) | 7 | 5 | 1 | 3
  Serotype 3: 5 days Post-Injection 1 | 1 | 0 | 0 | 0
  Serotype 3: 7 days Post-Injection 1: number analyzed (Participants) | 16 | 9 | 8 | 9
  Serotype 3: 7 days Post-Injection 1 | 5 | 2 | 1 | 4
  Serotype 3: 14 days Post-Injection 1: number analyzed (Participants) | 12 | 4 | 3 | 6
  Serotype 3: 14 days Post-Injection 1 | 1 | 1 | 0 | 1
  Serotype 3: 3 days Post-Injection 2: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 3: 3 days Post-Injection 2 |  |  |  | 0
  Serotype 3: 14 days Post-Injection 2: number analyzed (Participants) | 1 | 1 | 0 | 0
  Serotype 3: 14 days Post-Injection 2 | 0 | 0 |  |
  Serotype 3: 7 days Post-Injection 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Serotype 3: 7 days Post-Injection 3 | 1 |  |  |
  Serotype 4: 3 days Post-Injection 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 4: 3 days Post-Injection 1 |  |  |  | 0
  Serotype 4: 5 days Post-Injection 1: number analyzed (Participants) | 7 | 5 | 1 | 3
  Serotype 4: 5 days Post-Injection 1 | 6 | 3 | 1 | 2
  Serotype 4: 7 days Post-Injection 1: number analyzed (Participants) | 16 | 9 | 8 | 9
  Serotype 4: 7 days Post-Injection 1 | 13 | 7 | 5 | 7
  Serotype 4: 14 days Post-Injection 1: number analyzed (Participants) | 12 | 4 | 3 | 6
  Serotype 4: 14 days Post-Injection 1 | 8 | 2 | 2 | 4
  Serotype 4: 3 days Post-Injection 2: number analyzed (Participants) | 0 | 0 | 0 | 1
  Serotype 4: 3 days Post-Injection 2 |  |  |  | 0
  Serotype 4: 14 days Post-Injection 2: number analyzed (Participants) | 1 | 1 | 0 | 0
  Serotype 4: 14 days Post-Injection 2 | 0 | 0 |  |
  Serotype 4: 7 days Post-Injection 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Serotype 4: 7 days Post-Injection 3 | 0 |  |  |

7. Secondary Outcome: Geometric Means Titers of Antibodies Against Japanese Encephalitis - Groups 3 and 4
Description: GMTs of antibodies against JE were measured by JE micro neutralization assay. The LLOQ of the assay was a titer of 10 (1/dilution).
Time Frame: Pre-injection 1, and 28 days post-injection 1, 2 and 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 25 | 25
titers (1/dilution)
  Pre-injection 1: number analyzed (Participants) | 25 | 19
  Pre-injection 1 | NA [NA to NA] — Participants had a titer reported as < LLOQ. | 22.9 [12.7 to 41.0]
  28 days Post-injection 1: number analyzed (Participants) | 19 | 19
  28 days Post-injection 1 | 132.3 [48.4 to 361.9] | 620.9 [337.5 to 1142.3]
  28 days Post-injection 2: number analyzed (Participants) | 15 | 18
  28 days Post-injection 2 | 382.7 [134.7 to 1087.9] | 501.8 [253.0 to 995.5]
  28 days Post-injection 3: number analyzed (Participants) | 14 | 16
  28 days Post-injection 3 | 82.3 [40.3 to 167.9] | 157.4 [74.9 to 330.9]

8. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) pre-listed (i.e., solicited) in the electronic case report form (eCRF) and considered as related to vaccination. Solicited injection site reactions: pain, erythema, and swelling.
Time Frame: Within 7 days after any CYD dengue vaccine and/or JE vaccine
Population: Analysis was performed on safety analysis set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 24 | 15 | 22 | 19
Participants
  Injection site Pain | 7 | 6 | 3 | 6
  Injection site Erythema | 7 | 4 | 2 | 2
  Injection site Swelling | 3 | 2 | 0 | 1

9. Secondary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) pre-listed (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited systemic reactions: fever, headache, malaise, myalgia, and asthenia.
Time Frame: Within 14 days after any CYD dengue vaccine and/or JE vaccine
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- CYD Dengue and JE Vaccine: Group 4: Participants received 2 doses of JE (IXIARO) vaccines at 0 and 1 months; and 3 doses of CYD dengue vaccine at 7, 9 and 13 months, respectively.
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
Number analyzed (Participants) | 24 | 15 | 22 | 19
Participants
  Fever | 2 | 2 | 3 | 1
  Headache | 10 | 11 | 12 | 11
  Malaise | 9 | 10 | 11 | 6
  Myalgia | 8 | 6 | 10 | 7
  Asthenia | 6 | 7 | 7 | 3

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 up to 28 days after each dose of CYD dengue vaccine and/or JE vaccine. Solicited Reaction (SR) data were collected within 7 and 14 days after each and any vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 18 months for Groups 1, 2 and 3 and 19 months for Group 4).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was pre-listed (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and JE Vaccine : Group 3 | CYD Dengue and JE Vaccine: Group 4
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/25 | 0/15 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 18/25 | 15/15 | 17/25 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine: Group 1 (N=25) | CYD Dengue Vaccine: Group 2 (N=15) | CYD Dengue and JE Vaccine : Group 3 (N=25) | CYD Dengue and JE Vaccine: Group 4 (N=25)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine: Group 1 (N=25) | CYD Dengue Vaccine: Group 2 (N=15) | CYD Dengue and JE Vaccine : Group 3 (N=25) | CYD Dengue and JE Vaccine: Group 4 (N=25)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 6 (12) | 7 (11) | 7 (13) | 8 (14)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 7 (11) | 4 (6) | 2 (2) | 2 (2)
Injection site pain (General disorders) | 7 (8) | 6 (8) | 8 (13) | 13 (25)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 2 (3) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 9 (16) | 10 (12) | 11 (22) | 11 (23)
Pyrexia (General disorders) | 2 (3) | 2 (2) | 3 (3) | 2 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (7) | 2 (3) | 2 (2) | 6 (7)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 7 (7) | 3 (3) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (14) | 6 (11) | 10 (22) | 10 (22)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (27) | 13 (22) | 12 (37) | 14 (46)
Migraine (Nervous system disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications